CLINICAL TRIAL: NCT04367519
Title: Optic Nerve Sheath Diameter Versus Extra-vascular Lung Water Detected by Ultrasound in Volume Status Prediction in Severe Preeclampsia
Brief Title: Optic Nerve Sheath Diameter for Volume Status Prediction in Severe Preeclampsia
Status: Completed | Type: Observational
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Sherif M. S. Mowafy, Lecturer of anesthesia and surgical intensive care, Zagazig University
Other Study IDs: 6074-26-4-2020
Record Dates: First submitted 2020-04-26; First posted 2020-04-29 (Actual); Last update posted 2020-07-16 (Actual); Status verified 2020-07

CONDITIONS: Pre-Eclampsia
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Ultrasound measurement of Optic nerve sheath diameter — Ocular ultrasonography was performed with the patients placed in supine position with closed eyes. A layer of ultrasound gel was applied over the closed upper eyelid and the liner high frequency probe 7 - 12 MHz of SonoSite M-Turbo ultrasound machine was placed on the temporal area of the eyelid with the hand holding it resting on the forehead of the patient. The probe is then adjusted to a suitable angle in order to display the entry of the optic nerve into the globe. ONSD is then measured 3mm behind the globe in the transverse plane perpendicular to the optic nerve. For each eye one measurement will be made and the reported ONSD corresponds to the mean of the two values obtained for each patient. it was performed for all enrolled parturients within 24 hour before delivery and at 24 hour post-delivery.

SUMMARY:
A quick, non-invasive, bedside test to assess fluid status of patients with severe preeclampsia would be very helpful to ICU clinicians severe preeclampsia is associated with an increase in extravascular lung water (EVLW), which can be identified by lung ultrasound before appearance of clinical signs of pulmonary edema but this technique still requires several measurements and could be time consuming.

Optic ultrasound is also a safe and repeatable diagnostic tool, which is even quicker and simpler to perform than lung ultrasound. Increased ONSD is associated with increased ICP and it can indirectly reflect the state of intracranial edema that could be a part of generalized edema.

More data on the correlation between ONSD and markers of fluid status (EVLW by ultrasound) are needed before ONSD measurements can be recommended as a guide to fluid management in preeclampsia.

DETAILED DESCRIPTION:
Severe preeclampsia (PE) is a progressive multisystem pregnancy disorder. It is considered the second leading cause of maternal death worldwide. Usually, it is diagnosed by the new-onset hypertension and either proteinuria or end-organ dysfunction in the second half of pregnancy.

Acute Pulmonary edema is potentially lethal and is the most common cardiopulmonary complication of preeclampsia. thus, meticulous fluid management of these patients is crucial but it is often difficult because the underlying endothelial damage leads to water, electrolytes, and plasma leakage from the intravascular space which produce significant fluid shifts into the interstitial space resulting in peripheral and/or central (pulmonary and central nervous system) edema. Also, there is a potential for hypovolemia due to the depletion of intravascular volume. Under-resuscitation of preeclampsia patients impairs organ perfusion; while on the other hand fluid overload leads to tissue edema and aggravates pulmonary edema. Therefore, fluid administration must be assessed to preserve organ perfusion, while preventing lung congestion and pulmonary edema.

Early detection of lung congestion would allow early and optimal management of these patients. Lung ultrasound was reported as a useful diagnostic tool which could identify increased levels of extravascular lung water (EVLW) in severe PE before clinical signs of pulmonary edema appear. Consequently, lung ultrasound could guide fluid management and identify those in need for diuretic therapy among severe PE patients. Though it is considered accurate, safe, and non-invasive valuable tool, its use could be limited by the need to several measurements that could be time consuming.

Changes in the Optic Nerve Sheath Diameter (ONSD) detected by ultrasound are considered an important clinical and radiographic demonstration of increased intracranial pressure (ICP) which is one of the consequences of preeclampsia. Therefore, Increased ONSD can indirectly reflect the state of intracranial edema that could be a part of generalized edema.

On ultrasound the ONSD is measured 3 mm posterior to the globe for both eyes. A position of 3 mm behind the globe is recommended because the ultrasound contrast is greatest; the results are more reproducible and the normal optic nerve sheath measures up to 5.0 mm in diameter. An average ONSD greater than 5 mm is considered abnormal and elevated intracranial pressure should be suspected.

Chen et al., studied ONSD and the intravascular volume status of patients after cardiac surgery and found that changes in ONSD can dynamically reflect changes in volume status in patients with postoperative cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patient acceptance.
* Singleton Pregnant female complicated with severe preeclampsia
* Age 18-40 years old.
* Accepted mental state of the patient.

Exclusion Criteria:

* Patient refusal to participate to the study.
* Mild preeclampsia
* Uncooperative patient or altered sensorium
* Ocular wound
* Pneumonia
* Interstitial lung disease
* History of prior ocular trauma or surgery
* Preexisting heart disease
* Known pulmonary disorders.

Ages: 21 Years to 45 Years | Sex: Female
Age Groups: Adult
Study Population: Singleton Pregnant female complicated with severe preeclampsia. severe preeclampsia was determined by the presence of one or more of the following features using the American College of Obstetricians and Gynecologists severe features :
  * Systolic blood pressure ≥ 160 mmHg or diastolic blood pressure ≥ 110 mmHg on two occasions at least 4 hours apart
  * Thrombocytopenia (platelet count less than 100,000/L)
  * Impaired liver function indicated by elevated liver enzymes (to twice the upper limit normal concentration), and severe persistent right upper quadrant or epigastric pain not responding to medications and not explained by another diagnosis.
  * Renal insufficiency (serum creatinine concentration more than 1.1 mg/dL or doubling of the serum creatinine concentration in the absence of other renal disease)
  * Pulmonary edema
  * New-onset headache unresponsive to medications and not accounted for by alternative diagnoses
  * Visual disturbances
Sampling Method: Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-04-15 (Actual)

PRIMARY OUTCOMES:
the correlation of ONSD with EVLW | 24 hour
  Ultrasound assessment was performed for all enrolled preeclampsia patients within 24 hour before delivery and at 24 hour post-delivery.

CONTACTS AND LOCATIONS:
Overall Officials: Sherif M Mowafy, MD, Principal Investigator — Anesthesia and Surgical Intensive Care Department, Faculty of Medicine, Zagazig University; Mohamed I Elsayed, MD, Study Director — Anesthesia and Surgical Intensive Care Department, Faculty of Medicine, Zagazig University
Locations (1):
- Zagazig University Hospitals, Zagazig, Sharqia Province, Egypt

IPD SHARING:
Plan to Share IPD: Yes
all individual participant data that underlie results in the publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: the individual participant data and any additional supporting information will become available starting 6 months after publication.
Access Criteria: by contacting the study director

REFERENCES:
- [Background] Hariharan N, Shoemaker A, Wagner S. Pathophysiology of hypertension in preeclampsia. Microvasc Res. 2017 Jan;109:34-37. doi: 10.1016/j.mvr.2016.10.002. Epub 2016 Oct 26. No abstract available. PMID 27793558
- [Background] Melchiorre K, Sharma R, Thilaganathan B. Cardiovascular implications in preeclampsia: an overview. Circulation. 2014 Aug 19;130(8):703-14. doi: 10.1161/CIRCULATIONAHA.113.003664. No abstract available. PMID 25135127
- [Background] Dennis AT, Solnordal CB. Acute pulmonary oedema in pregnant women. Anaesthesia. 2012 Jun;67(6):646-59. doi: 10.1111/j.1365-2044.2012.07055.x. Epub 2012 Mar 15. PMID 22420683
- [Background] Chaiworapongsa T, Chaemsaithong P, Yeo L, Romero R. Pre-eclampsia part 1: current understanding of its pathophysiology. Nat Rev Nephrol. 2014 Aug;10(8):466-80. doi: 10.1038/nrneph.2014.102. Epub 2014 Jul 8. PMID 25003615
- [Background] Pretorius T, van Rensburg G, Dyer RA, Biccard BM. The influence of fluid management on outcomes in preeclampsia: a systematic review and meta-analysis. Int J Obstet Anesth. 2018 May;34:85-95. doi: 10.1016/j.ijoa.2017.12.004. Epub 2017 Dec 20. PMID 29398426
- [Background] Zieleskiewicz L, Contargyris C, Brun C, Touret M, Vellin A, Antonini F, Muller L, Bretelle F, Martin C, Leone M. Lung ultrasound predicts interstitial syndrome and hemodynamic profile in parturients with severe preeclampsia. Anesthesiology. 2014 Apr;120(4):906-14. doi: 10.1097/ALN.0000000000000102. PMID 24694847
- [Background] Shyamsundar M, Attwood B, Keating L, Walden AP. Clinical review: the role of ultrasound in estimating extra-vascular lung water. Crit Care. 2013 Sep 13;17(5):237. doi: 10.1186/cc12710. PMID 24041261
- [Background] Ambrozic J, Brzan Simenc G, Prokselj K, Tul N, Cvijic M, Lucovnik M. Lung and cardiac ultrasound for hemodynamic monitoring of patients with severe pre-eclampsia. Ultrasound Obstet Gynecol. 2017 Jan;49(1):104-109. doi: 10.1002/uog.17331. Epub 2016 Dec 1. PMID 27736042
- [Background] Sekhon MS, Griesdale DE, Robba C, McGlashan N, Needham E, Walland K, Shook AC, Smielewski P, Czosnyka M, Gupta AK, Menon DK. Optic nerve sheath diameter on computed tomography is correlated with simultaneously measured intracranial pressure in patients with severe traumatic brain injury. Intensive Care Med. 2014 Sep;40(9):1267-74. doi: 10.1007/s00134-014-3392-7. Epub 2014 Jul 18. PMID 25034476
- [Background] Pordeus ACB, Katz L, Soares MC, Maia SB, Amorim MMR. Acute pulmonary edema in an obstetric intensive care unit: A case series study. Medicine (Baltimore). 2018 Jul;97(28):e11508. doi: 10.1097/MD.0000000000011508. PMID 29995818
- [Background] ACOG Practice Bulletin No. 202: Gestational Hypertension and Preeclampsia. Obstet Gynecol. 2019 Jan;133(1):1. doi: 10.1097/AOG.0000000000003018. PMID 30575675
- [Background] Volpicelli G, Elbarbary M, Blaivas M, Lichtenstein DA, Mathis G, Kirkpatrick AW, Melniker L, Gargani L, Noble VE, Via G, Dean A, Tsung JW, Soldati G, Copetti R, Bouhemad B, Reissig A, Agricola E, Rouby JJ, Arbelot C, Liteplo A, Sargsyan A, Silva F, Hoppmann R, Breitkreutz R, Seibel A, Neri L, Storti E, Petrovic T; International Liaison Committee on Lung Ultrasound (ILC-LUS) for International Consensus Conference on Lung Ultrasound (ICC-LUS). International evidence-based recommendations for point-of-care lung ultrasound. Intensive Care Med. 2012 Apr;38(4):577-91. doi: 10.1007/s00134-012-2513-4. Epub 2012 Mar 6. PMID 22392031
- [Background] Picano E, Pellikka PA. Ultrasound of extravascular lung water: a new standard for pulmonary congestion. Eur Heart J. 2016 Jul 14;37(27):2097-104. doi: 10.1093/eurheartj/ehw164. Epub 2016 May 12. PMID 27174289
- [Background] Dubost C, Le Gouez A, Jouffroy V, Roger-Christoph S, Benhamou D, Mercier FJ, Geeraerts T. Optic nerve sheath diameter used as ultrasonographic assessment of the incidence of raised intracranial pressure in preeclampsia: a pilot study. Anesthesiology. 2012 May;116(5):1066-71. doi: 10.1097/ALN.0b013e318246ea1a. PMID 22258019